CLINICAL TRIAL: NCT06409052
Title: Endometrial Cancer, Risk Factors and Prevention Strategies: Perspectives of Patients and At-Risk Women
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0443; NCI-2023-08979 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Qualitative interviews — Interviews will be conducted for approximately 45-60 minutes

SUMMARY:
To learn more about women's attitudes toward and knowledge about endometrial cancer and options that might decrease the risk of developing

DETAILED DESCRIPTION:
To obtain pilot data regarding women's attitudes and perspectives about endometrial cancer and potential endometrial cancer prevention strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Women who present to MD Anderson Cancer Center including MDA Houston Area Locations with a diagnosis of endometrial cancer
2. Women who present to MD Anderson Cancer Center including MDA Houston Area Locations with a diagnosis of abnormal uterine bleeding or endometrial hyperplasia
3. Women without a diagnosis of endometrial cancer or endometrial hyperplasia
4. Women must be at least 18 years or age
5. Women must be able to read, write, and speak English
6. Women must be willing and able to provide written informed consent

Exclusion Criteria:

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women with or without a diagnosis of endometrial cancer or endometrial hyperplasia
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2026-08-03 (Estimated); Study Completion 2026-08-03 (Estimated)

PRIMARY OUTCOMES:
Patient education | Through study completion; an average of 1 year.
  To build a patient tool for educating and empowering women to make informed decisions about endometrial cancer prevention strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Larissa Meyer, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org